CLINICAL TRIAL: NCT04909151
Title: The Effect of Robot-assisted Gait Training on Gait Ability in Children With Cerebral Palsy
Brief Title: The Effect of Robot-assisted Gait Training on Gait Ability in Children With Cerebral Palsy Through Changing Gait Speed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, Principal Investigator, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-1040781-A-N-012021050HR
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy; Gait Disorders, Neurologic; Bilateral Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic | interventions — Walking Speed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot-assisted gait training with walking speed of 0.5km/h (Experimental)
  Interventions: Device: Robot-assisted gait training (walking speed: 0.5km/h)
- Robot-assisted gait training with walking speed of 0.8km/h (Experimental)
  Interventions: Device: Robot-assisted gait training (walking speed: 0.8km/h)
- Robot-assisted gait training with walking speed of 1.1km/h (Experimental)
  Interventions: Device: Robot-assisted gait training (walking speed: 1.1km/h)

INTERVENTIONS:
Device: Robot-assisted gait training (walking speed: 0.5km/h) — Robot-assisted gait training RAGT, WALKBOT-G, is a walking training equipment that can reproduce natural motions by adjusting the leg length and adjusting the motion with the actuator of the ankle joint.
  Arms: Robot-assisted gait training with walking speed of 0.5km/h
Device: Robot-assisted gait training (walking speed: 0.8km/h) — Robot-assisted gait training RAGT, WALKBOT-G, is a walking training equipment that can reproduce natural motions by adjusting the leg length and adjusting the motion with the actuator of the ankle joint.
  Arms: Robot-assisted gait training with walking speed of 0.8km/h
Device: Robot-assisted gait training (walking speed: 1.1km/h) — Robot-assisted gait training RAGT, WALKBOT-G, is a walking training equipment that can reproduce natural motions by adjusting the leg length and adjusting the motion with the actuator of the ankle joint.
  Arms: Robot-assisted gait training with walking speed of 1.1km/h

SUMMARY:
Robot-assisted gait training (RAGT) improves the gait ability of children with cerebral palsy, and can provide treatment plans and guidelines through changed records of various gait variables. There is a lack of concrete explanations or arguments for gait speed, weight support ratio, support force, joint angle, etc. that can be set in the RAGT system, and intervention intensity for an appropriate intervention program has not been presented. Therefore, in this study, we would like to suggest clinically effective interventions for children with cerebral palsy in the second stage of the gross motor function classification system (GMFCS) by identifying gait variables according to differences in gait speed during RAGT.

ELIGIBILITY:
Inclusion Criteria:

* Patients 4-12 years old diagnosed with cerebral palsy
* Children who have not received botulinum toxin treatment or surgery within 3 months
* Children in stage 2 of the gross motor function system
* Children who can express pain, fear, or discomfort on their own

Exclusion Criteria:

* Severe lower extremity contracture and fracture
* Bone instability
* Osteoporosis
* Severe bones grow disproportionately
* Unhealed skin lesions on the lower extremities (thromboembolic disease)
* Thromboembolic disease
* Cardiovascular instability
* Mild scoliosis with a Cobb's angle of more than 20 degrees

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Gait ability | Change from baseline gait ability at 6 weeks
  Gait ability is evaluated using the Zebris FDM-Treadmill. When the participants walks on the treadmill, the foot pressure is recorded at a rate of 120 Hz. The input pressure signal is displayed as a 2D/3D graph including the center of pressure while standing or walking, and the spatiotemporal measurements are displayed.

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Geon Park, Ph.D candidate, Principal Investigator — The Wells Neuro Pain Clinic
Locations (1):
- Pajucity convalescent Hospital, Paju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
I plan to decide after the study is over.